CLINICAL TRIAL: NCT04190758
Title: GOTHA - The Early Arthritis and Psoriasis Study of Region Västra Götaland, Sweden
Acronym: GOTHA
Status: Enrolling by invitation | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: VastraGotaland record 273244
Record Dates: First submitted 2019-12-04; First posted 2019-12-09 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis; Arthritis; Psoriasis; Cardiovascular Diseases; Obesity; Lung Diseases
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Arthritis; Psoriasis; Cardiovascular Diseases; Obesity; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma will be sampled at each study visit. DNA and RNA tubes and fecal samples will be collected at baseline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Patients with rheumatoid arthritis (RA): Patients with RA meeting the classification criteria of American College of Rheumatology (ACR) and/or European League Against Rheumatism (EULAR) från 2010.
  Interventions: Other: Care as usual
- Patients with psoriatic arthritis (PsA): Patients with PsA meeting the classification criteria of Classification for Psoriatic Arthritis (CASPAR).
  Interventions: Other: Care as usual
- Patients with undifferentiated arthritis: Defined as a patients with a clear arthritis, but not meeting with established classifications criteria of any now known rheumatic disease.
  Interventions: Other: Care as usual
- Patients with psoriasis: Patients with psoriasis diagnosed at a dermatology department. The patients should not have any history of joint complaints with a duration of more than 6 weeks.
  Interventions: Other: Care as usual
- General population controls: General population controls retrieved from the Population Register, matched for age, sex and residence of living to the included patients.

INTERVENTIONS:
Other: Care as usual — No intervention will be given. The study will follow the effects of care as usual.
  Groups: Patients with psoriasis; Patients with psoriatic arthritis (PsA); Patients with rheumatoid arthritis (RA); Patients with undifferentiated arthritis

SUMMARY:
GÖTHA- The early arthritis and psoriasis study of Region Västra Götaland, Sweden - is a longitudinal observational study, which will prospectively and in parallel follow patients with newly diagnosed rheumatoid arthritis (RA, N=1000), psoriatic arthritis (PsA, N=500) and undifferentiated arthritis (N=100), together with patients with psoriasis (N=500). The study will also recruit healthy controls from the general population (N=3000).

The aims of the study are to define predictors for disease course and severity, treatment response, comorbidities, health related quality of life (HRQoL) and health economy.

The study is a collaboration between the department of Rheumatology and the department of Dermatology at Sahlgrenska University Hospital in Gothenburg, and the departments of Rheumatology at the hospitals of Alingsås, Borås, Uddevalla and Skövde, in the west of Sweden.

All patients with newly diagnosed RA, PsA and undifferentiated arthritis at the Rheumatology centers are eligible for inclusion. Patients with psoriasis will be recruited from the Department of dermatology at Sahlgrenska University Hospital.

The patients will be examined at baseline and at one, three, five and ten years. The assessments will include physical examination with evaluation of joints, entheses and skin and validated questionnaires regarding medical history, comorbidities, lifestyle, disease activity, bodily function, socioeconomic factors and HRQoL. Blood samples will be collected. The patients with arthritis will also undergo radiography of the lung, hands and feet, and Cone Beam Computed Tomography (CBCT) of hands and feet.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rheumatoid arthritis (RA) meeting the classification criteria of American College of Rheumatology (ACR) and/or European League Against Rheumatism (EULAR) från 2010
* Patients with psoriatic arthritis (PsA) meeting the classification criteria of Classification for Psoriatic Arthritis (CASPAR) PsA
* Patients with undifferentiated arthritis defined as a patients with a clear arthritis, but not meeting with established classifications criteria of any now known rheumatic disease
* Patients with psoriasis diagnosed at a dermatology department. The patients should not have any history of joint complaints with a duration of more than 6 weeks
* General population controls, matched for age, sex and residence of living to the included patients.

Exclusion Criteria:

* Inability to follow study protocol
* Swedish language difficulties
* Having other concomitant rheumatic diagnose (Sjögrens syndrome is not an exclusion criteria)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients at any of the involved rheumatology clinics with newly diagnosed RA, PsA or undifferentiated arthritis meeting the study criteria are eligible for inclusion.
  Consecutive sampling
  Patients with psoriasis diagnosed at a dermatology clinic. Consecutive sampling
Sampling Method: Non-Probability Sample
Enrollment: 5100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2039-12-31 (Estimated); Study Completion 2069-12-21 (Estimated)

PRIMARY OUTCOMES:
Disease activity | 12 months
  Disease Activity Score using 28 joint counts (DAS28) score range 0-9.07

CONTACTS AND LOCATIONS:
Overall Officials: Eva Klingberg, Assoc. Prof, Principal Investigator — Dep of Rheumatology and Inflammation research, University of Gothenburg, Sweden; Inger Gjertsson, Prof, Principal Investigator — Dep of Rheumatology and Inflammation research, University of Gothenburg, Sweden
Locations (1):
- Clinical Rheumatology Research Center (CRRC), Department of Rheumatology, Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided